CLINICAL TRIAL: NCT05557578
Title: Tislelizumab Combined with GEMOX (GOT) Applied As Neoadjuvant Regimen for Patients of Resectable Intrahepatic Cholangiocarcinoma with High-risk Factors of Recurrence: a Single Arm, Single Center, Prospective, Explorative Clinical Trail.
Brief Title: GOT Applied As Neoadjuvant Regimen for Patients of Resectable ICC with High-risk Factors of Recurrence
Acronym: GOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yuhua Zhang, MD, Vice director of Hepatobiliary and Pancreatic Surgery, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhangYH
Record Dates: First submitted 2022-09-19; First posted 2022-09-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Tislelizumab; Gemcitabine; Oxaliplatin; cholangiocarcinoma; Neoadjuvant
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Clinical Protocols; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Patients of Resectable ICC With High-risk Factors of Recurrence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Tislelizumab combined with GEMOX (GOT) regimen
  Interventions: Drug: Tislelizumab combined with GEMOX (GOT) regimen

INTERVENTIONS:
Drug: Tislelizumab combined with GEMOX (GOT) regimen — Tislelizumab 200mg on day 1；Gemcitabine 1000mg/m2 on day 1、8；Oxaliplatin 135mg/m2 on day 1；cycle 3 weeks
  Other Names: Gemcitabine; Oxaliplatin

SUMMARY:
Intrahepatic cholangiocarcinoma (ICC) arises from the epithelial cells of bile ducts and occurs proximal to the segmental biliary ducts. ICC is highly aggressive, long-term survival only can be achieved in patients with R0 surgical resection. Large diameter of tumor, multiple tumors, preoperative carbohydrate antigen(CA)19-9 elevated, tumors invaded adjacent blood vessels and preoperative radiology hints suspected regional lymph node metastasis were considered as high-risk factors of recurrence in the previous study. Chemotherapy can trigger antigen release and induces strong anti-tumor effects of T cells due to cytotoxic cell death. Immune checkpoint inhibitors can relieve tumor immunosuppressive microenvironment. Hence, we aim to investigate objective response rate and R0 resection rate and survival rate of patients with high-risk factors of recurrence who receives Tislelizumab combined with GEMOX regimen(GOT) as a neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 yo;
2. Patients of Pathological confirmed intrahepatic cholangiocarcinoma who has never received systemic therapy including chemotherapy, immunotherapy, target therapy and other anti-cancer therapy;
3. Patients of resectable ICC with high risk recurrent factors:

   ①Maximum diameter greater than 5cm or multiple tumors.

   ②Preoperative CA19-9 greater than 200 Unit(U)/mL

   ③Tumors invaded adjacent blood vessels

   ④Preoperative radiology hints suspected regional lymph node metastasis.

   ⑤Tumor tissues confirmed by CT or MRI, at least one measurable lesion exists according to RECIST v1.1.
4. Eastern Cooperative Oncology Group(ECOG)-Performance status(PS) score is 0 before first drug administration;
5. Child-Pugh classification is class A;
6. Estimated overall survival is greater than 16 weeks;
7. The level of organ function meets the criteria and can tolerate surgery before the first treatment. Main organs meet the criteria as below:

   haemoglobin≥90g/L，Neutrophil count≥1.5×10⁹/L，Platelet count≥100×10⁹/L；Aspartate or alanine aminotransferase≤5 upper limits of normal(ULN），alkaline phosphatase≤2.5 ULN，Serum albumin≥30g/L；serum creatinine<1.5 ULN；International normalized ratios（INR）≤2 or Prothrombin time（PT）exceed ULN≤6s；Creatinine clearance≥60 mL/min.
8. Male and female subjects with potential fertility had to agree to the use of effective contraceptive methods throughout the study period；
9. Sign an informed consent form agreeing to provide previously preserved specimens of tumor tissue or fresh detection of tumor lesions.

Exclusion Criteria:

1. Patient with non-intrahepatic cholangiocarcinoma；
2. Anti-cancer therapy or surgery such as radiotherapy, radiofrequency ablation, interventions in 28 days prior to the first dose of the study (except for previous non-tumor-related surgeries and diagnostic biopsies)；
3. Distant metastasis；
4. hepatitis B virus (HBV) DNA>2000 copies/ml, hepatitis C virus (HCV) RNA>1000;
5. Long-term glucocorticoid users require long-term systemic hormones (equivalent to >10 mg Prednisone/day) or any other form of immunosuppressive therapy；
6. Clinically significant bleeding or bleeding tendencies within 3 months prior to enrollment or on thrombolytic or anticoagulant therapy；
7. Patients with complete bowel obstruction and incomplete intestinal obstruction that require treatment, but patients who have been relieved of obstruction by ostomy or stent placement can be enrolled；
8. Active severe clinical infections (> grade 2, NCI-CTCAE version 5.0), including active TB; Have a history of active TB infection at least 1 year before enrolment, have not received regular anti-tuberculosis (TB) treatment or are still active; active, known or suspected autoimmune disease;
9. Uncontrolled diabetes mellitus (fasting blood glucose ≥10 mmol/L), severe lung disease (eg, acute lung disease, pulmonary fibrosis that affects lung function, interstitial lung disease). except for recovered radiation pneumonia);
10. Clinically significant cardiovascular diseases; With hypertension, antihypertensive drugs cannot be well controlled (systolic blood pressure≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
11. Patient who are receiving renal replacement therapy；
12. History of other malignancies in the last 5 years. With the exception of carcinoma of the skin basal cells that have been cured or carcinoma in situ in the cervix;
13. Others situations are not expected to tolerate surgical treatment；
14. People with allergic reactions to any component of the drug under study;
15. There are other unsuitable candidates for clinical trials, such as alcohol dependence, mental illness, pregnancy (or lactation).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 6 cycle treatment (each cycle is 21 days), an average of 18 weeks.
  The proportion of patients who achieved complete response (CR) and partial response(PR) after GOT regimen neoadjuvant treatment according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
R0 resection rate | Up to pathological report come out, an average of 20 weeks.
  The proportion of patients who achieved pathological negative surgical margin after GOT regimen neoadjuvant treatment.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 6 cycle treatment (each cycle is 21 days), an average of 18 weeks.
  The proportion of patients who achieved complete response (CR), partial response (PR) and stable disease (SD) after GOT regimen neoadjuvant treatment according to RECIST v1.1.
Recurrence free survival | From date when patients are received radical resection until the date of first documented recurrence radiologically, assessed at least 12 months.
  The time between the date of patients underwent radical resection and the date of radiographic recurrence as defined by RECIST1.1.
Overall survival | From date when patients are received radical resection until the date of death from any cause, assessed at least 12 months.
  The time between the date of patients underwent radical resection and death from any cause.

OTHER OUTCOMES:
Time to response (TTR) | From date of received first treatment to first achieved complete or partial response, up to 18 weeks.
  The time between the date of patients received first treatment and the date of first documented complete or partial response.
Time to operation (TTO) | From date of received first treatment to date of surgery, an average of 20 weeks.
  The time between the date of patients received first treatment and the date of patients received operation.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhua - Zhang, M.D., Study Chair — Zhejiang Cancer Hospital
Locations (2):
- China (2):
  - 1# Banshan East Rd. Zhejiang cancer hospital, Hangzhou, Zhejiang
  - Jia Wu, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided